CLINICAL TRIAL: NCT02666495
Title: Individual Schema-mode Therapy for Anorexia Nervosa: a Pilot Case Series
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015/0228
Record Dates: First submitted 2016-01-25; First posted 2016-01-28 (Estimated); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Anorexia Nervosa
Keywords: Schema Therapy
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Psychological Therapy - Schema Therapy — Psychological treatment using individual Schema-Mode Therapy for Anorexia Nervosa (iST-AN). A 60 session protocol will be used over an 18 month period, moving flexibly through five phases of treatment, guided by the psychological formulation: phase 1 - assessment, engagement & stabilisation; phase 2 - developing trust & understanding; phase 3 - developing awareness & acceptance; phase 4 - testing change & strengthening the healthy mode; phase 5 - consolidating change. A follow-up period of 6 months, with 5 further monthly sessions, will promote self-efficacy and further consolidate change. A total treatment package of 65 sessions will be offered, over 24 months.

SUMMARY:
A reliably effective treatment model for anorexia nervosa is yet to emerge. Recent clinical trials of psychological therapies over 20-30 sessions, have shown modest benefits. There is therefore a need to test new treatments to find more effective treatments. Clinical trials of Schema Therapy have shown low rates of dropout, which is often a problem in the treatment of anorexia nervosa. Treatment with Schema Therapy, for significantly longer than 20-30 sessions, has been shown to be effective for other complex mental health problems.This pilot study is therefore designed to pilot the use of individual Schema Therapy for people with Anorexia Nervosa (iST-AN). This study is a case series pilot study. The study will answer the principal research question: Does individual Schema mode Therapy, adapted for eating disorders, have the potential to improve symptoms, quality of life and weight in people with moderate-severe anorexia nervosa? It will also address secondary research questions: Can people with moderate-severe anorexia nervosa be recruited to, and kept engaged in, a study of iST-AN treatment? What is the ideal length of iST-AN treatment? What is the relationship between self-criticism, body shame, or unhelpful psychological 'modes' and clinical outcome? Fifteen people with moderate-severe Anorexia Nervosa will be recruited from referrals to a specialist eating disorders outpatient service. The study will deliver 65 sessions of Schema Therapy for anorexia nervosa (iST-AN), over a 24 month period, alongside any additional medical or dietetic management required. Standard outcome measures will be collected at 6 month intervals. The research team have expertise in eating disorders research, schema therapy for severe anorexia nervosa and are all members of the local clinical service. The study will take place over a 3 year period.

DETAILED DESCRIPTION:
Aims & Hypotheses

The aims of this pilot case series of individual Schema-mode Therapy for Anorexia Nervosa (iST-AN) are:

1. To test the potential efficacy of iST-AN treatment, including

   1. exploring optimal length of treatment
   2. refining the iST-AN treatment manual
2. To test recruitment and retention in iST-AN treatment
3. To explore hypotheses relating to self-criticism, body shame & change in strength of modes.

We anticipate that treatment with iST-AN will result in adequate recruitment and a high level of retention in treatment. We hypothesise that treatment with iST-AN will result in significant change in eating disorder symptoms, quality of life (QoL) and body mass index (BMI). We hypothesise that improved symptoms, QoL and BMI will correlate with reduced self-criticism, reduced body shame and reduced strength of maladaptive coping modes.

Methods Population & Recruitment Our intention is to recruit a broadly representative population of adults with moderate-severe, treatment resistant or co-morbid Anorexia Nervosa (AN). Outpatients will be recruited from The Cullen Centre, Edinburgh, Scotland. Recruitment will occur from routine referrals and we anticipate recruiting 10-15 cases over a 12 month period.

Assessment Procedures

Stage 1 - Screening:

Any patient referred to the service who may fulfil the inclusion criteria, is eligible for screening, including those on waiting lists at the start of the recruitment period. Every patient identified for screening will be allocated a unique identification number prior to screening, by the data manager. Screening will be carried out by the study therapist by telephone or face-to-face, to supplement the referral information. This will be guided by the study screening questionnaire. Self-report BMI, age, and history of previous schema therapy treatment, will be established using the screening questionnaire. If screen positive, the potential participant is offered an eligibility assessment appointment during the screening call, and sent a patient information sheet about the study and schema therapy, along with a letter confirming the assessment appointment.

Stage 2 - Eligibility and clinical assessment appointment:

The eligibility assessment will be combined with a standard clinical assessment, carried out by the study therapist and colleagues, according to local protocols. The study therapist will complete the eligibility questionnaire and assessments. The Eating Disorders Examination (edition 17.0D), the 5 diagnostic items, will be used to make valid DSM-V underweight eating disorder diagnoses. The MINI structured diagnostic interview and the self-report Personality Belief Questionnaire (PBQ) will be used to define co-morbidity for psychotic disorders, alcohol or drug dependence or misuse, personality disorder, obsessive-compulsive disorder, other anxiety disorders and depressive disorders. A standard clinical assessment will screen for possible learning disability or Autistic Spectrum Disorder. The potential participant is given an opportunity at this appointment to ask any questions about the study.

Following this appointment the eligibility information is reviewed. Participants are contacted by phone within one week to offer entry to the study or advice regarding the local treatment service if they are ineligible for the study or choose to not participate. This will be confirmed by letter.

Stage 3 - Informed consent & baseline assessments appointment:

Any further questions will be addressed at this appointment prior to obtaining informed consent. Demographic and treatment history information will be gathered by the study therapist using a bespoke study questionnaire. This includes assessment of: duration of eating disorder; previous therapy for eating disorder; lowest ever BMI; relationship status; employment status; and current medication. The participant will also be given time at this appointment to complete the battery of baseline outcome questionnaires, with the therapist available for clarification if required. The option of completing the questionnaires at home will be available if preferred.

Treatment Patients will be treated using a manualised but flexible treatment protocol. Engaging people with anorexia nervosa in treatment is notoriously difficult. The value people with anorexia nervosa attach to their disorder, combined with difficulties trusting others and over-controlling behaviour, means that a flexible individualised treatment approach is likely to enhance engagement. A 60 session protocol will be used over an 18 month period, moving flexibly through five phases of treatment, guided by the psychological formulation: phase 1 - assessment, engagement & stabilisation; phase 2 - developing trust & understanding; phase 3 - developing awareness & acceptance; phase 4 - testing change & strengthening the healthy mode; phase 5 - consolidating change. A follow-up period of 6 months, with 5 further monthly sessions, will promote self-efficacy and further consolidate change. A total treatment package of 65 sessions will be offered, over 24 months. Some therapy sessions will be audio recorded for quality assurance and supervision purposes.

Medical and psychiatric risk management will continue as per local service protocols. Should inpatient care be required, patients will be retained in the trial if an admission is limited to less than 8 weeks, with admissions recorded for reporting in results. Patients who lose capacity to consent to participation in the trial, who are admitted for longer than 8 weeks or require use of the mental health act, will be withdrawn from the trial and further treatment will be determined by local protocols. Treatment with medication and dietetic treatment will continue as per local service protocols and recorded for reporting in results. These measures will ensure any significant additional treatment beyond iST-AN is reported clearly within our results and that no patient is denied any locally available adjunctive treatment alongside the psychological therapy.

Data Management and Analysis An assistant psychologist from Edinburgh eating disorder services will be the data manager, with the support of the Scottish Mental Health Research Network (SMHRN). A unique identification number will be allocated sequentially to each patient entering the screening process. All outcome measures will be collected at baseline, 6, 12, 18 and 24 months, with the exception of the SMI, to be collected at baseline and 24 months only, due to the length of this questionnaire.

Questionnaire packs will be provided electronically by the data manager, alongside a system of reminders sent two weeks prior to the set data point. Participants will be encouraged to complete questionnaires on paper at the clinic, but will have the option to complete these at home or online at www.surveymonkey.com. The Treating clinicians will ensure completion of outcome measures and passing this information to the data manager. The anonymised data with a unique identification number, will be managed and stored on the password-secured IT systems of the University of Edinburgh.

Analyses will be conducted using the Statistical Package for the Social Sciences, version 21 (SPSS v21). We will describe the numbers of patients screened, recruited and retained in treatment. Using the intention to treat principle, repeated measure linear mixed-model analyses (LMM) will be used to assess efficacy on each of our measures of outcome: symptoms, weight gain and quality of life. The pattern of change will be examined to explore whether a 65 session treatment package appears too long or too short. We will also explore our hypotheses that reduced self-criticism, reduced body shame and reduced strength of maladaptive coping modes will be correlated with positive outcomes, using multivariate analysis of variance (MANOVA).

Timeline

1. Ethics approval: Feb-Mar 2015
2. Local R&D approval: Mar-Apr 2015
3. Recruitment: Jan 2016- Jan 2017
4. Completion of data collection: Jan 2019
5. Completion of analysis: May 2019
6. Grant submission for multi-centre RCT of iST-AN: By Dec 2018
7. Submission for publication: By Dec 2018

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of AN or other DSM-V underweight eating disorder diagnosis AND
2. 18 yrs or over AND
3. Moderate-severe, treatment resistant, comorbid, or chronic 3.1. BMI 13-15 OR 3.2. BMI 15-17.5 and ≥ 1 previous treatment episode for eating disorder OR 3.3. BMI 15-17.5 and a personality disorder diagnosis OR 3.4. BMI 15-17.5 and duration of eating disorder of > 10 yrs

Exclusion Criteria:

1. Diagnosis of psychotic disorder
2. Diagnosis of alcohol or drug dependence
3. Diagnosis of learning disability or autistic spectrum disorder
4. English language skills not adequate for therapy
5. Previous treatment with Schema Mode Therapy
6. Unable to make realistic commitment to attend weekly appointments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2015-01-25 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Eating Disorders Examination questionnaire (EDE-Q) | 6 monthly
  A validated self-report measure of eating disorder symtpoms.

SECONDARY OUTCOMES:
Body Mass INdex (BMI) | 6 monthly
  standardised method of calculation of weight relative to height.
WHO-QoL (bref) | 6 monthly
  A validated self-report measure of quality of life
Symptom Check List - 90 | 6 monthly
  A validated self-report measure of general psychiatric symptoms.
Global Assessment of Functioning (GAF) | 6 monthly
  A clinician rated measure of general symptoms and funcctioning

OTHER OUTCOMES:
Forms of Self-Criticism/Self-Reassuring scale (FSCRS) | 6 monthy
  A validated self-report measure of self-criticism
Body shame items of the Experiences of Shame Scale (ESS) | 6 monthly
  A validated self-report measure of body-shame
Schema Mode Inventory (SMI) | baseline and 24 months
  A validated self-report measure of psychological self-states

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Edinburgh Hospital, Edinburgh, United Kingdom